CLINICAL TRIAL: NCT00916422
Title: Clinical, Multi-centre,Randomized, Double-blind, Placebo-controlled Subcutaneous Immunotherapy Trial With Depigmented, Polymerised Extract of Phleum Pratense Pollen on Patients With Hypersensitivity to Grass Pollen
Brief Title: Subcutaneous Immunotherapy Treatment for Patients With Hypersensitivity to Grass Pollen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-005868-10
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2012-08

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Immunotherapy; Allergoid; Depigmented; Polymerized; Allergen-extract; Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Allergens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depigoid Phleum pratense 1000DPP/Ml (Experimental): Depigmented and Polymerized Allergen extract of Phleum Pratense.Subcutaneous Immunotherapy in an up-dosing cluster regimen for 4 weeks, followed by monthly injections for 2 years.
  Interventions: Biological: Allergen extract (Phleum pratense)
- 2 (Placebo Comparator): Placebo. Dosing regimen: An up-dosing cluster regimen for 4 weeks, followed by monthly injections for 2 years
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Allergen extract (Phleum pratense) — Subcutaneous immunotherapy with modified extract of Phleum pratense. A subcutaneous monthly treatment.
  Arms: Depigoid Phleum pratense 1000DPP/Ml
Biological: Placebo — Subcutaneous monthly treatment
  Arms: 2

SUMMARY:
The objective of this trial is to assess the clinical efficacy of the modified extract (depigmented and polymerised with glutaraldehyde)of the subcutaneous injection of Phleum pratense pollen in the treatment of patients affected by allergic rhinitis/ rhinoconjunctivitis ( with or without episodic asthma) induced by hypersensitivity to grass pollen, evaluating the Score regarding Symptoms and consumption of the medication.

DETAILED DESCRIPTION:
Immunotherapy is a specific treatment for allergic diseases. Unlike conventional pharmacological treatment, immunotherapy is the only treatment that could modify the natural course of allergic disease. This is a prospective double-blind placebo controlled study with two arms of treatment in an up-dosing cluster regimen for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, signed by the subject.
* Clinical History of moderate to severe rhinitis/rhinoconjunctivitis lasting for at least 2 consecutive years, with or without episodic asthma, caused by allergy to grass pollen.
* Patient of both gender aged from 18 up to 55
* Symptoms that coincide with allergy to grass pollen
* Sensitivity to grass pollen, diagnosed through a positive skin reaction to Phleum pratense: Positive prick test and /or Specific IgE to P.pratense >0,7KU/L Patients included must be mono-sensitised or, in the case of poly-sensitisation, sensitivity to p.pratense pollen should be considered as the only relevant aspect of their condition from the clinical standpoint.
* Patients who are able to comply with the dose regime

Exclusion Criteria:

* Patient with mild Rhinitis/rhinoconjunctivitis
* Relevant sensitivity to another perennial allergen
* Use of immunotherapy during the last four years
* Treatment with B. Blocking agents
* Patient suffering from some pathology in which adrenalin was contraindicated
* Subject suffers from a serious medical condition, which would interference the treatment and follow up of the subject in the study
* Subject suffers from autoimmune disease(thyroiditis, lupus, etc.)
* Conditions in which the patient can not offer full co-operation and significant psychiatric disorders.
* Intolerance to aspirin
* Pregnant women or with pregnancy risk and breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2008-06; Primary Completion 2013-01 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Symptoms and medication score recorded by subjects | 2 year

SECONDARY OUTCOMES:
Nasal provocation test, Dose-response skin prick test, Rhinoconjunctivitis Quality of life questionnaire, visual scales, asthma symptom scores, medication scores, adverse event and severity adverse event, unplanned health care resource utilization | 2

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Sanchez, Principal Investigator — Hospital Río Carrión
Locations (23):
- Hungary (4):
  - Fövarosi Önkormányzat Szent János Kórháza és Észak-budai Egyesített, Budapest, Budapest
  - AEK Jarobetegszakrendelo Intézet Pulmonologia, Budapest, Budapest
  - Selye jános Kórhaz-Rendelöintézet Tüdögondozó Intézet, Komárom, Komárom
  - Karolina Kórhaz Rendelöintézet Tüdögondozó, Mosonmagyaróvár, Mosonmagyaróvár
- Spain (19):
  - Hospital Universitario de Getafe, Madrid, Madrid
  - H. Río Carrión, Palencia, Palencia
  - Hospital Ntra. Sra de Sonsoles, Ávila
  - Hospital de Llerena, Badajoz
  - Hospital Militar de Burgos, Burgos
  - Hospital de Coria, Cáceres
  - Hospital Ntra. Sra. de la Montaña, Cáceres
  - Hospital Ciudad Real, Ciudad Real
  - Hospital San Juan de Dios, León
  - Hospital Virgen Blanca, León
  - Hospital San Millan, Logroño
  - Hospital de Merida, Mérida
  - Clinica Universitaria de Navarra, Navarra
  - Hospital del Bierzo, Ponferrada
  - Hospital Santa Barbara, Puertollano
  - Hospital de Santa Barbara, Soria
  - Hospital Universitario del Río Hortega, Valladolid
  - Hospital Clinico Lozano Blesa, Zaragoza
  - Hospital la Maz, Zaragoza